CLINICAL TRIAL: NCT01503606
Title: Duration of Antibiotics Treatment With Cefazolin and Clarithromycin in Women With Preterm Premature Rupture of Membrane, Phase III Study.
Brief Title: Duration of Antibiotics Treatment With Cefazolin and Clarithromycin in Women With Preterm Premature Rupture of Membrane
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Oh Soo Young, Associate professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2011-07-005
Record Dates: First submitted 2011-12-25; First posted 2012-01-04 (Estimated); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Preterm Premature Rupture of Membrane
Keywords: preterm premature rupture of membrane; antibiotics; duration; cefazolin; clarithromycin
MeSH Terms: conditions — Preterm Premature Rupture of the Membranes | interventions — Cefazolin; Clarithromycin

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- one-week treatment group (Active Comparator): Cefazolin 1.0gm IVs q 12 hours plus clarithromycin 500mg po bid after randomization for one week
  Interventions: Drug: Cefazolin; Drug: Clarithromycin
- until-delivery treatment group (Active Comparator): Cefazolin 1.0gm IVs q 12 hours plus clarithromycin 500mg po bid after randomization until delivery
  Interventions: Drug: Cefazolin; Drug: Clarithromycin

INTERVENTIONS:
Drug: Cefazolin — Cefazolin 1.0gm IVs q 12 hours after randomization for one week
  Arms: one-week treatment group
Drug: Clarithromycin — clarithromycin 500mg po bid after randomization for one week
  Arms: one-week treatment group
Drug: Cefazolin — Cefazolin 1.0gm IVs q 12 hours after randomization until delivery
  Arms: until-delivery treatment group
Drug: Clarithromycin — clarithromycin 500mg po bid after randomization until delivery
  Arms: until-delivery treatment group

SUMMARY:
The purpose of this study is to compare the neonatal outcome and infant neurologic outcome whose mother were treated with cefazolin plus clarithromycin for one week or until delivery after preterm premature rupture of membrane.

ELIGIBILITY:
Inclusion Criteria:

* preterm premature rupture of membrane(PPROM), PA 22+0~34+0wks
* ROM <72 hrs before randomization
* cervical dilatation <3cm
* uterine contraction less than 4 times per 1 hr

Exclusion Criteria:

* Major fetal malformation
* Rupture of the membrane >72hrs before randomization
* Vaginal bleeding
* IIOC (incompetent internal os of cervix)
* Placenta previa
* Gestational diabetes or overt diabetes
* Hypertensive disorders in pregnancy
* Liver cirrhosis
* Acute renal failure

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2011-10; Primary Completion 2020-12 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Neonatal composite morbidity | Participants will be followed for duration of hospital day after delivery, an expected average of 8 weeks
  1. respiratory distress syndrome(RDS)
  2. bronchopulmonary dysplasia(BPD)
  3. intraventricular hemorrhage(IVH,≥grade 3)
  4. retinopathy of prematurity(ROP,≥grade 3)
  5. necrotizing enterocolitis(NEC,≥stage 2)
  6. proven neonatal sepsis

SECONDARY OUTCOMES:
infantile neurologic outcome | at 6 months and 1 year of corrected age
  The outcome will be evaluated in five sub-domains (development, neurologic examination, Bayley Scales of Infant Development-II, vision, and hearing). The final outcome scale was divided into normal, mild, moderate, and severe disability

CONTACTS AND LOCATIONS:
Overall Officials: Soo-young Oh, MD, PhD, Principal Investigator — Samsung Medical Center, Sungkyunkwan University School of Medicine
Locations (1):
- Samsung Medical center, Sungkyunkwan University School of Medicine, Seoul, South Korea

REFERENCES:
- [Derived] Sung JH, Kim JH, Kim Y, Choi YS, Hong S, Choi SJ, Kim JS, Roh CR, Oh SY. A randomized clinical trial of antibiotic treatment duration in preterm pre-labor rupture of membranes: 7 days vs until delivery. Am J Obstet Gynecol MFM. 2023 Apr;5(4):100886. doi: 10.1016/j.ajogmf.2023.100886. Epub 2023 Feb 4. PMID 36746334